CLINICAL TRIAL: NCT02288624
Title: A Randomized, Double Blind and Crossover Study Investigating the Effect of Whole Versus Processed Orange Consumption on Satiety in Healthy Volunteers
Brief Title: The Effects of Whole Versus Processed Orange Consumption on Satiety
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Reading (Other)
Collaborators: PepsiCo Global R&D (Industry)
Responsible Party: Principal Investigator, Jeremy Paul Edward Spencer, Professor of nutritional medicine, University of Reading
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: UOR-0002
Record Dates: First submitted 2014-01-16; First posted 2014-11-11 (Estimated); Last update posted 2014-11-11 (Estimated); Status verified 2014-11

CONDITIONS: Satiety Response

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Control (Placebo Comparator): Water control (240 ml)
  Interventions: Dietary Supplement: Processed orange juice
- Orange Juice (Experimental): Orange juice, 240 ml. Commercial orange juice
  Interventions: Dietary Supplement: Processed orange juice
- Whole orange (Experimental): Whole orange, 240 ml. Whole orange, blended to include all edible orange material.
  Interventions: Dietary Supplement: Processed orange juice
- processed orange juice (Experimental): Processed orange juice, 240 ml. Experimental orange juice processing
  Interventions: Dietary Supplement: Processed orange juice

INTERVENTIONS:
Dietary Supplement: Processed orange juice — 3 different formulation of edible orange drinks

SUMMARY:
This is a human dietary intervention study that is randomized and crossover in design with 4 treatment arms consisting of control, orange juice,whole orange, and processed whole orange to investigate the satiety effects of the treatments in healthy volunteers. Self reported hunger and fullness scores by Visual Analogue Scale (VAS) form were collected at different time points prior to and post consumption of each treatment.

DETAILED DESCRIPTION:
This is a human dietary intervention study that is randomized and crossover in design with 4 treatment arms consisting of control, orange juice,whole orange, and processed whole orange to investigate the satiety effects of the treatments in healthy volunteers. Self reported hunger and fullness scores by Visual Analogue Scale (VAS) form were collected at different time points prior to and post consumption of each treatment.

ELIGIBILITY:
Inclusion Criteria:

* Gender: male or female(postmenopausal women only)
* Age at start of the study: males ≥ 21and ≤ 65 years and females ≥ 50 and ≤ 65 years
* Body Mass Index (BMI) ≥ 18.5 and ≤ 27 kg/m2
* Apparently healthy: measured by questionnaire, no reported current or previous metabolic diseases or chronic gastrointestinal disorders
* Reported dietary habits: no medically prescribed diet, no slimming diet, used to eating 3 meals a day
* Reported intense sporting activities ≤ 10h/w
* Reported alcohol consumption ≤21 units/w
* Informed consent signed
* Recruitment form filled out

Exclusion Criteria:

* Smoking
* Dislike, allergy or intolerance to test products
* Possible eating disorder (measured by SCOFF questionnaire score >1)
* Eating habits questionnaire score >14
* Reported medical treatment that may affect eating habits/satiety
* Pre menopausal women

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2012-04; Primary Completion 2013-04 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Self reported hunger and fullness score by Visual Analogue Scale | baseline to 2 hours

SECONDARY OUTCOMES:
Overall liking by '9 point hedonic scale' | baseline to 2 hours

CONTACTS AND LOCATIONS:
Overall Officials: Jeremy P Spencer, PhD, Principal Investigator — University of Reading
Locations (1):
- Hugh Sinclair Unit of Human Nutrition, Reading, Berkshire, United Kingdom